CLINICAL TRIAL: NCT00921960
Title: St. Vincent's Screening To Prevent Heart Failure (STOP-HF) Study Using Natriuretic Peptides to Identify and Prevent Progression of Left Ventricular Dysfunction in Community Based, Asymptomatic, At-risk Individuals.
Brief Title: St. Vincent's Screening To Prevent Heart Failure Study
Acronym: STOP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's University Hospital, Ireland (Other)
Collaborators: University College Dublin (Other); Crofton Cardiac Centre, Dublin (Unknown); The Heartbeat Trust (Other)
Responsible Party: Principal Investigator, Mark Ledwidge, Research Director, Heart Failure Unit St Vincent's University Hospital, St Vincent's University Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SVUH - HFU - 020
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Left Ventricular Dysfunction; Myocardial Infarction; Hypertension; Diabetes; Obesity
Keywords: Left ventricular dysfunction; Left ventricular systolic dysfunction; Left ventricular diastolic dysfunction; Myocardial Infarction; Hypertension; Diabetes; Obesity; Dyslipidaemia; Heart Failure; Prevention; Screening; Cardiovascular Risk Factors; Echocardiography; Natriuretic Peptides
MeSH Terms: conditions — Ventricular Dysfunction, Left; Myocardial Infarction; Hypertension; Diabetes Mellitus; Obesity; Dyslipidemias; Heart Failure | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual Care will involve ongoing management from the general practitioner, nurse-led assessment of cardiovascular risk at the general practice and referral to specialist services as deemed necessary.
- Intervention (Other): Intervention Care is defined as a collaborative cardiovascular management between primary care and specialist hospital based services. This will involve natriuretic peptide guided evaluation of LVD and follow-up as appropriate
  Interventions: Other: Intervention Care

INTERVENTIONS:
Other: Intervention Care — Intervention Care is defined as a collaborative cardiovascular management between primary care and specialist hospital based services. This will involve natriuretic peptide guided evaluation of LVD and follow-up as appropriate - for example including echocardiographic assessment of left ventricular systolic dysfunction and appropriate pharmacotherapy.
  Other Names: Screening; Health services delivery intervention
  Arms: Intervention

SUMMARY:
The STOP-HF study is a prospective, randomized, controlled trial recruiting asymptomatic individuals with risk factors for left ventricular dysfunction from 50 primary care clinics in Dublin and south east Ireland. It is designed to determine whether using natriuretic peptide measurement as a screening tool following a general cardiovascular risk factor screen will reduce the prevalence and severity of ventricular dysfunction in conjunction with specialist follow-up at St. Vincent's University Hospital.

DETAILED DESCRIPTION:
A large proportion of the population has substantial left ventricular dysfunction (LVD) and do not have symptoms (Stage B heart failure). For many of these patients, if identified and treated appropriately, it is possible to prevent the subsequent development of heart failure (HF). Although the current gold standard for detection of LVD is echocardiography, it is expensive and impractical for mass screening.

Natriuretic peptides are attractive candidates for screening populations for asymptomatic LVD particularly because of high negative predictive values. Furthermore, some studies have shown that, in the right setting, screening with natriuretic peptides might prove cost effective in combination with echocardiography for patients with elevated levels.

However, in common with many accepted screening strategies, there are no randomised studies which show that screening the population with natriuretic peptides for asymptomatic LVF alters the natural history of the condition.

From a large, community based cardiovascular risk screening programme including more than 13,000 patients, patients in the catchment area of St Vincent's University Hospital are invited to participate in the STOP-HF study. The objective of this work is to determine whether or not using natriuretic peptide screening in conjunction with specialist follow-up will reduce the prevalence and severity of LVD in a well-defined, at-risk, primary care population. It also aims to: evaluate the natural history of natriuretic peptides over time in this population; to clarify optimal screening cut-offs for the detection of LVD; to evaluate the clinical, pharmacological, biochemical, genetic and proteomic determinants of natriuretic peptides in this setting; to determine whether the clinical benefits of the STOP HF screening programme, if any, are cost effective.

The study design is prospective, randomised and parallel group.

The primary endpoint is the prevalence and severity LVD after 5 years of follow up. Secondary endpoints include: the natural history of natriuretic peptides; the relationship between natriuretic peptides and severity of LVD, death, hospital admissions; clinical, demographic, biochemical, pharmacological, genomic, proteomic, metabolomic determinants of natriuretic peptides; screening cost-effectiveness.

Participants who fulfill entry criteria at baseline will sign an informed consent and will be randomised onto the Usual Care or Intervention Care arm of the study. Usual care is defined as continued management of the patient by the primary care services using standard risk factor monitoring and intervention strategies. Intervention Care is defined as a collaborative cardiovascular management between primary care and specialist hospital based services. All participants will receive an intensive education session from a cardiovascular nurse on their risk factors and advice on healthy dietary and lifestyle habits.

There will be 2 years of enrollment with annual review and 5 years of follow-up to the primary endpoint. Permission has been received to extend the follow up period to 10 years. Regardless of randomisation, all patients receive full clinical and laboratory assessment at baseline and on completion of the STOP HF study (year 5). Additionally, all participants will receive echocardiography assessment during and at the conclusion of the study.

Data collection:

Data will be collected on all participants regarding their medical history and current medications. The source of data collection will be from medical records kept at the primary care practices and from patient interview. All participants will receive a booklet in which they will be asked to record any visits to their primary care practitioner, alterations in medications, new diagnoses and hospital admissions. Local hospital discharge records will be screened to detect any events throughout the course of the study.

Clinical Assessment:

At annual intervals, the cardiovascular research nurse will conduct clinical assessments on all participants including weight, abdominal girth measurement, blood pressure (triplicate measurements while lying in supine position), heart rate and observe for evidence of limb oedema. The nurse will also question the participants to investigate for symptoms of dyspnoea, angina, palpitations, orthopnoea, palpitations and fatigue.

Blood sampling and handling:

Peripheral venous blood samples will be drawn on all participants at annual intervals. Samples to assess natriuretic peptides will be drawn into vacutainers containing EDTA and samples to assess renal function, collagen turnover and lipid profile will be collected in vacutainers containing lithium heparin. BNP and Lipid profile assessment will be analysed using point of care meters, Biosite (Triage, USA) and Cholestech respectively. Each of the remaining samples will be centrifuged for 10 minutes and the serum will be then aliquoted and stored at -80°C before analysis of biochemical, genomic, proteomic and metabolomic markers.

Echocardiographic Doppler analysis:

Two-dimensional echocardiographic imaging, targeted M-mode and Doppler ultrasound measurements will be obtained in each patient. M-mode measurements are taken according to the guidelines laid down by the American Society of Echocardiography. All echocardiographic data will represent the mean of 3 measurements on different cardiac cycles. It is the aim of the STOP HF investigators that a single observer will conduct all measurements, recording archive images in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 Years of age
* with risk factors for LVD including:

  * hypertension (medicated for ≥ 1 month)
  * hypercholesterolemia
  * obesity
  * coronary artery disease (confirmed by angiography)
  * diabetes mellitus
  * arrhythmia
  * valvular abnormalities

Exclusion Criteria:

* failure or unwilling to provide informed consent
* known ventricular dysfunction (confirmed by angiography or echocardiography)
* previous documented episode of heart failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1378 (Estimated)
Dates: Start 2005-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of LVD | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M McDonald, MD, Principal Investigator — St Vincent's University Hospital, Ireland; Mark T Ledwidge, PhD, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St Vincent's University Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Sweeney C, Pharithi RB, Kerr B, Ryan C, Ryan F, Collins L, Halley C, Barrett M, Watson CJ, McDonald K, Ledwidge M. NT-proBNP/BNP ratio for prognostication in European Caucasian patients enrolled in a heart failure prevention programme. ESC Heart Fail. 2021 Dec;8(6):5081-5091. doi: 10.1002/ehf2.13576. Epub 2021 Sep 29. PMID 34586748
- [Derived] Watson C, Spiers JP, Waterstone M, Russell-Hallinan A, Gallagher J, McDonald K, Ryan C, Gilmer J, Ledwidge M. Investigation of association of genetic variant rs3918242 of matrix metalloproteinase-9 with hypertension, myocardial infarction and progression of ventricular dysfunction in Irish Caucasian patients with diabetes: a report from the STOP-HF follow-up programme. BMC Cardiovasc Disord. 2021 Feb 12;21(1):87. doi: 10.1186/s12872-021-01860-7. PMID 33579197
- [Derived] Ledwidge MT, O'Connell E, Gallagher J, Tilson L, James S, Voon V, Bermingham M, Tallon E, Watson C, O'Hanlon R, Barry M, McDonald K. Cost-effectiveness of natriuretic peptide-based screening and collaborative care: a report from the STOP-HF (St Vincent's Screening TO Prevent Heart Failure) study. Eur J Heart Fail. 2015 Jul;17(7):672-9. doi: 10.1002/ejhf.286. PMID 26139583
- [Derived] Ledwidge M, Gallagher J, Conlon C, Tallon E, O'Connell E, Dawkins I, Watson C, O'Hanlon R, Bermingham M, Patle A, Badabhagni MR, Murtagh G, Voon V, Tilson L, Barry M, McDonald L, Maurer B, McDonald K. Natriuretic peptide-based screening and collaborative care for heart failure: the STOP-HF randomized trial. JAMA. 2013 Jul 3;310(1):66-74. doi: 10.1001/jama.2013.7588. PMID 23821090
- [Derived] Bermingham M, Hayden J, Dawkins I, Miwa S, Gibson D, McDonald K, Ledwidge M. Prospective analysis of LDL-C goal achievement and self-reported medication adherence among statin users in primary care. Clin Ther. 2011 Sep;33(9):1180-9. doi: 10.1016/j.clinthera.2011.07.007. Epub 2011 Aug 12. PMID 21840055